CLINICAL TRIAL: NCT06537583
Title: The Efficacy and Safety of Low-Level Tragus Stimulation on Heart Rate Variability, Neutrophil-Lymphocyte Ratio, and Major Adverse Cardiovascular Events in Patients With ST-Segment Elevation Myocardial Infarction
Brief Title: The Efficacy and Safety of Low-Level Tragus Stimulation on Heart Rate Variability, Neutrophil-Lymphocyte Ratio, and Major Adverse Cardiovascular Events in Patients With ST-Segment Elevation Myocardial Infarction (TESLA-STEMI)
Acronym: TESLA-STEMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Diponegoro (Other)
Responsible Party: Principal Investigator, Sodiqur Rifqi, Principal Investigator; Former of Head of Department of Cardiovascular Medicine Faculty of Medicine Universitas Diponegoro, Universitas Diponegoro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Undip
Record Dates: First submitted 2024-07-24; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: ST segment elevation myocardial infarction; Low level tragus stimulation; Heart rate variability; Neutrophil-lymphocyte ratio; Major adverse cardiovascular events
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant will not know either they include in treatment or control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Level Tragus Stimulation Group (Experimental): Participant will undergo low level tragus stimulation using Parasym Device
  Interventions: Device: Parasym Neuromodulation Device (Treatment Group); Device: Parasym Neuromodulation Device (Sham Group)
- Sham Control Group (Sham Comparator): Participant will have Parasym Device implanted in their tragus without any active stimulation from the device
  Interventions: Device: Parasym Neuromodulation Device (Treatment Group); Device: Parasym Neuromodulation Device (Sham Group)

INTERVENTIONS:
Device: Parasym Neuromodulation Device (Treatment Group) — Participant will undergo stimulation in their left tragus for 60 minutes by using Parasym device
Device: Parasym Neuromodulation Device (Sham Group) — Participant will undergo implantation of Parasym device lead in their left tragus but without any stimulation for 60 minutes

SUMMARY:
The goal of this clinical trial is to learn the effect of low level tragus stimulation (LLTS) on heart rate variability (HRV), neutrophil-lymphocyte ratio, and major adverse cardiovascular events in patient with ST-segment Elevation Myocardial Infarction (STEMI). It will also learn about the safety of LLTS in such setting. The main questions, it aims to answer are compared with sham control:

1. Does LLTS could alter low frequency/high frequency ratio in patients with STEMI?
2. Does LLTS could alter neutrophil-lymphocyte ratio in patients with STEMI?
3. Does LLTS could decrease mortality in patients with STEMI?
4. Does LLTS could decrease reinfarction event in patients with STEMI?
5. Does LLTS could decrease stroke event in patients with STEMI?
6. Does LLTS could decrease lethal arrhythmia event in patients with STEMI?
7. Does LLTS could decrease acute lung oedema event in patients with STEMI?
8. Does LLTS could decrease cardiogenic shock event in patients with STEMI?

Researchers will compare LLTS to sham LLTS control to see if LLTS have benefit in participants with STEMI participants will divided into two group i.e. treatment group vs control (sham/placebo) group, then both of them:

1. Undergo laboratory examination before Primary Percutaneous Coronary Intervention (PPCI)
2. Undergo HRV measurement using WeCardio device before Primary Percutaneous Coronary Intervention (PPCI)
3. Undergo LLTS (treatment group will have stimulation) for 60 minutes, however, sham control will not have stimulation, before PPCI
4. Undergo PPCI
5. Undergo laboratory examination after Primary Percutaneous Coronary Intervention (PPCI)
6. Undergo HRV measurement using WeCardio device after Primary Percutaneous Coronary Intervention (PPCI)

ELIGIBILITY:
Inclusion Criteria:

* Onset STEMI less than 12 hours
* Participant agreed to be included in this study
* Killip class I - II on presentation
* SBP >90 mmHg and/or MAP >65 mmHg
* Sinus rhtyhm

Exclusion Criteria:

* History of myocardial infarction, stroke, heart failure with reduce ejection fraction, chronic total occlussion on prior coronary angiography, chronic kidney disease (eGFR < 30) or on hemodyalisis, malignancy, hematology disease, autoimmune, or other chronic diseases
* On permanent pacemaker
* Acute infection
* Pregnant woman

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events | During hospitalization around up to 1 weeks
  Consist of mortality, reinfarction, stroke, lethal arrhtyhmia, acute lung oedema, cardiogenic shock

SECONDARY OUTCOMES:
Heart Rate Variability | Before and After LLTS and Primary PCI (approximately within 24 to 48 hours after PPCI)
  Heart Rate Variability measurement by using WeCardio device
Neutrophil-Lymphocyte Ratio | Before and After LLTS and Primary PCI (approximately within 24 to 48 hours after PPCI)
  Neutrophil-Lymphocyte Ratio from laboratory findings

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Kariadi Central General Hospital, Semarang, Central of Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu L, Huang B, Po SS, Tan T, Wang M, Zhou L, Meng G, Yuan S, Zhou X, Li X, Wang Z, Wang S, Jiang H. Low-Level Tragus Stimulation for the Treatment of Ischemia and Reperfusion Injury in Patients With ST-Segment Elevation Myocardial Infarction: A Proof-of-Concept Study. JACC Cardiovasc Interv. 2017 Aug 14;10(15):1511-1520. doi: 10.1016/j.jcin.2017.04.036. PMID 28797427
- [Background] Redgrave J, Day D, Leung H, Laud PJ, Ali A, Lindert R, Majid A. Safety and tolerability of Transcutaneous Vagus Nerve stimulation in humans; a systematic review. Brain Stimul. 2018 Nov-Dec;11(6):1225-1238. doi: 10.1016/j.brs.2018.08.010. Epub 2018 Aug 23. PMID 30217648